CLINICAL TRIAL: NCT02066961
Title: A Prospective, Longitudinal, Multinational, Observational Study to Describe Patterns of Care and Outcomes of Men Who Are at High Risk for Poor Clinical Outcomes After Experiencing Biochemical Failure Following Definitive Prostate Cancer Therapy, Men With Castration-Resistant Prostate Cancer and Men With Metastatic Prostate Cancer at Initial Diagnosis
Brief Title: A Study to Describe Patterns of Care and Outcomes of Men Who Are at High Risk After Experiencing Biochemical Failure Following Definitive Prostate Cancer Therapy, Men With Castration-resistant Prostate Cancer and Men With Metastatic Prostate Cancer
Acronym: ASPIRE-PCa
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ONC-MA-1001
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Prostate Cancer
Keywords: metastatic prostate cancer; castration-resistant prostate cancer; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Subjects with biochemical failure experience after primary treatment and have high-risk disease
- Cohort 2: Subjects with a medical diagnosis of castration-resistant prostate cancer
- Cohort 3: Subjects with an initial diagnosis of metastatic prostate cancer

SUMMARY:
The purpose of this study is to describe patterns in disease management and to describe clinical outcomes, as well as to identify factors influencing physician treatment decisions including reason(s) for treatment choices and trigger(s) for treatment changes and to document healthcare resource utilization used to manage treatment-related complications.

DETAILED DESCRIPTION:
Each subject will be followed from the time of enrollment for a minimum of 3 years and a maximum of up to 6 years or until death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate adenocarcinoma
* Will receive a new intervention at the time of study entry, for the treatment of:

  * Biochemical failure after initial curative-intent surgery (radical prostatectomy) or radiotherapy (external-beam radiation therapy, brachytherapy, or both) and a PSA doubling time of one year or less or a confirmed PSA of ≥ 50 ng/mL (2 consecutive values) within 6 months prior to study entry; or
  * Castration-resistant prostate cancer; or
  * Metastatic prostate cancer at initial diagnosis of prostate cancer

Exclusion Criteria:

* Prior treatment of metastatic castration-resistant prostate cancer with systemic chemotherapy
* Life expectancy of <1 year due to comorbidities

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from the offices of either a medical oncologist, radiation oncologist, uro-oncologist, urologist, surgeon, or primary care physician.
Sampling Method: Non-Probability Sample
Enrollment: 1533 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Patterns of disease management | up to 72 months
  Description of disease assessment methods, physician referral patterns and treatments
Clinical outcomes | up to 72 months
  Evidence of disease progression and development of symptomatic disease

SECONDARY OUTCOMES:
Factors influencing physician treatment decisions | up to 72 months
  Reason/s for treatment choices and trigger/s for treatment changes
Documentation of healthcare resource utilization used to manage treatment-related complications | up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (78):
- Algeria (2):
  - Site, Algiers
  - Site, Blida
- Argentina (3):
  - Site, Buenos Aires
  - Site, La Pampa
  - Site, Paraje Cabal
- Australia (5):
  - Site, Port Macquarie, New South Wales
  - Site, Tweed Heads, New South Wales
  - Site, Kurralta Park, South Australia
  - Site, Parkville, Victoria
  - Site, Richmond, Victoria
- Site, Vienna, Austria
- Brazil (7):
  - Site, Belo Horizonte, Minas Gerais
  - Site, Ijuí, Rio Grande do Sul
  - Site, Passo Fundo, Rio Grande do Sul
  - Site, Porto Alegre, Rio Grande do Sul
  - Site, São Paulo, São Paulo
  - Site, Caxias do Sul
  - Site, Santo André
- Canada (2):
  - Site, Granby, Quebec
  - Site, Québec, Quebec
- Colombia (2):
  - Site, Bogotá, DC
  - Site, Cali
- Site, Cairo, Egypt
- France (7):
  - Site, Besançon
  - Site, Lille
  - Site, Nîmes
  - Site, Pierre-Bénite
  - Site, Poitiers
  - Site, Saint-Mandé
  - Site, Suresnes
- Germany (7):
  - Site, Berlin
  - Site, Freiburg im Breisgau
  - Site, Hamburg
  - Site, Jena
  - Site, Nürtingen
  - Site, Rostock
  - Site, Ulm
- Site, Jakarta, Indonesia
- Israel (2):
  - Site, Beer Ya'akov, Zerifin
  - Site, Haifa
- Italy (4):
  - Site, Brescia
  - Site, Cremona
  - Site, Milan
  - Site, Orbassano
- Site, Beirut, BA, Lebanon
- Site, Durango, Mexico
- Netherlands (2):
  - Site, Amsterdam
  - Site, Nijmegen
- New Zealand (3):
  - Site, Hamilton, Waikato Region
  - Site, Christchurch
  - Site, Tauranga
- Site, Muscat, Oman
- Peru (2):
  - Site, Miraflores, Lima region
  - Site, Lima
- Philippines (3):
  - Site, Makati
  - Site, Pasig
  - Site, San Juan City
- Site, Riyadh, Saudi Arabia
- Site, Singapore, Singapore
- South Korea (5):
  - Site, Anyang
  - Site, Busan
  - Site, Incheon
  - Site, Seoul
  - Site, Suwon
- Spain (3):
  - Site, Vall d'Hebron 119-129, Barcelona
  - Site, Madrid
  - Site, Sabadell
- Taiwan (4):
  - Site, Guishan Township, Taoyuan County
  - Site, Kaohsiung City
  - Site, Taichung
  - Site, Taipei
- Thailand (3):
  - Site, Bangkok
  - Site, Phayathai
  - Site, Songkhla
- United Kingdom (4):
  - Site, Hull
  - Site, London
  - Site, Newcastle upon Tyne
  - Site, Sunderland

IPD SHARING:
Plan to Share IPD: Undecided